CLINICAL TRIAL: NCT05027932
Title: Randomized, Double-Blinded, Placebo-Controlled, Phase 1 Study of the Safety and Immunogenicity of BPL-1357, A BPL-Inactivated, Whole-Virus, Universal Influenza Vaccine
Brief Title: Safety and Immunogenicity of BPL-1357, A BPL-Inactivated, Whole-Virus, Universal Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10000320; 000320-I (Other: NIH)
Record Dates: First submitted 2021-08-28; First posted 2021-08-31 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Influenza
Keywords: Flu; Immunity; Virology; Investigational; Healthy Volunteer
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): 15 participants receiving IM BPL1357 & IN Placebo
  Interventions: Other: IN Placebo; Drug: BPL-1357
- Group B (Experimental): 15 participants receiving IN BPL1357 & IM Placebo
  Interventions: Other: IM Placebo; Drug: BPL-1357
- Group C (Sham Comparator): 15 participants receiving IM and IN placebo
  Interventions: Other: IN Placebo; Other: IM Placebo

INTERVENTIONS:
Other: IN Placebo — The placebo is normal saline in two syringes administered IN.
  Arms: Group A; Group C
Other: IM Placebo — The placebo is normal saline in a syringe administered IM.
  Arms: Group B; Group C
Drug: BPL-1357 — BPL-1357 contains 4 whole inactivated avian influenza viruses: A /Environment /Maryland/261/2006 H7N3, A/Mallard /Maryland/802/2007 H5N1, A/Pintail/Ohio /339/1987 H3N8, and A/Mallard/Ohio /265/1987 H1N9. It is administered either IM or IN depending on the assigned treatment group.
  Arms: Group A; Group B

SUMMARY:
Background:

Influenza (flu) is a virus that infects people of all ages. Some people may have mild flu symptoms. Others may get very sick and even die from the flu. Flu vaccines help protect people against the flu, but if the flu strains in the vaccine are not a good match with the strains circulating in the community, the vaccine is not as effective. Researchers want to make flu vaccines that protect against changing flu strains.

Objective:

To test if a new flu vaccine is safe and if it creates an immune response.

Eligibility:

Healthy adults ages 18-55 who do not smoke and have not received a flu vaccine in the 8 weeks prior or a COVID-19 vaccine in the 4 weeks prior to enrollment.

Design:

Participants will be screened on a separate protocol.

Participants will have 9 visits over 7 months. They will get a combination of study vaccine and/or placebo, both as a shot in the arm and as a spray into the nose, at 2 visits. For 7 days after getting the vaccines, they will take their temperature and complete online surveys at home to record any symptoms.

At each visit, participants will have a physical exam and medical history. They will give blood and urine samples. They will have nasal testing. For this, a thin absorptive strip will be inserted into their nostril for 1 minute to collect mucus. At some visits, the inside of their nose will be wiped with a small brush to collect cells. For this, their nostril will be numbed to make it more comfortable. Some blood and nasal samples will be used for genetic testing. Participants who get flu-like symptoms during the study will be asked to collect nasal samples at home and send these samples back to NIH to test if they actually have the flu.

DETAILED DESCRIPTION:
Study Description: This is a randomized, double-blinded, placebo-controlled, single-center, phase 1 clinical trial of beta-propiolactone (BPL)- inactivated quadruple influenza virus cocktail vaccine (BPL-1357) administered intramuscularly (IM) or intranasally (IN) in 2 doses 28 days apart. Participants will be randomized to one of three groups for treatment assignment. The primary hypothesis is that IN and IM BPL-1357 will be well tolerated.

Objectives:

Primary Objective:

1. To assess the safety of BPL-1357 given IM or IN, compared to placebo.

Secondary Objective:

1. To further assess the safety of BPL-1357 given IM or IN, compared to placebo.
2. To assess the immunogenicity of BPL-1357 given IM or IN, compared to placebo.

Tertiary Objective:

1. To characterize the systemic and mucosal humoral immune responses induced by BPL-1357 given IM or IN, compared to placebo.
2. To further characterize the immune response induced by BPL-1357 given IM or IN through variable, diversity, and joining (VDJ) gene repertoire analysis, cytokine analysis, cytometry, transcriptomics, and assessment of T-cell responses.
3. To assess the rates of influenza disease among groups given IM or IN BPL-1357 compared to placebo.

Endpoints:

Primary Endpoints:

1. Type and severity (by grading) of adverse events (AEs) through vaccine 2 (V2) day 28 (D28) [28 days after vaccine dose 2].
2. Type of serious adverse events (SAEs) through V2D28 [28 days after vaccine dose 2].

Secondary Endpoints:

1. Safety

   1. Type and severity (by grading) of AEs through V2D182 [182 days after vaccine dose 2].
   2. Type of SAEs through V2D182 [182 days after vaccine dose 2].
2. Immunogenicity

   1. Antibodies against H1, H3, H5, and H7 head and stalk as measured by hemagglutination inhibition (HAI) or enzyme-linked immunosorbent assay (ELISA) from blood and mucosal samples at V2D28.
   2. Antibodies against N1, N3, N8, and N9 as measured by neuraminidase inhibition (NAI) or ELISA from blood and mucosal samples at V2D28.

Tertiary Endpoints:

1. Additional antibody titer characterization via:

   1. Antibodies against H1, H3, H5, and H7 head and stalk as measured by HAI or ELISA from blood and mucosal samples at V1D7, V1D14, V1D28, V2D7, V2D14, V2D56, and V2D182.
   2. Antibodies against N1, N3, N8, and N9 as measured by NAI or ELISA from blood and mucosal samples at V1D7, V1D14, V1D28, V2D7, V2D14, V2D56, and V2D182.
2. Additional immune response characterization via:

   1. VDJ gene repertoire analysis.
   2. Cytokine analysis.
   3. Flow cytometric phenotyping of lymphocytes.
   4. Transcriptomic gene expression.
   5. T-cell responses.
3. Influenza disease

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* 18 and <= 55 years of age.

  * Non-smoker (tobacco and cannabis) and does not use vape or e-cigarette products.
  * Has not received influenza vaccination of any type in the 8 weeks prior to enrollment and willing to not receive influenza vaccination of any type until after the V2D56 visit. Participants who enroll in our study will be informed of the Centers for Disease Control and Prevention (CDC) recommendation to receive seasonal influenza vaccination annually.
  * Has not received Coronavirus Disease 19 (COVID-19) vaccination of any type in the 4 weeks prior to enrollment and willing to not receive COVID-19 vaccination of any type until after the V2D28 visit. Participants who enroll in our study who are interested in getting a COVID-19 vaccination will be counselled to receive it prior to enrolling into our study.
  * A female participant is eligible for this study if she is not pregnant or breastfeeding and meets one of the following criteria, beginning at least 4 weeks prior to enrollment through the end of the study period (V2D182):

    * Is infertile, including postmenopausal status (as defined by no menses for >= 1 year) or history of hysterectomy or bilateral oophorectomy.
    * Agrees to practice abstinence.
    * Agrees that, with heterosexual intercourse with a fertile male partner, she will use an acceptable form of contraception and her male partner will use a condom with spermicide. Acceptable effective methods of female contraception include the following: bilateral tubal ligation, implant of levonorgestrel, injectable progestogen, intrauterine device, oral contraceptive pills, and diaphragm with spermicide.
  * Able to provide informed consent.
  * Able to speak English.
  * Human immunodeficiency virus (HIV) uninfected with a negative test within 60 days of enrollment.
  * Does not use IN medications (including but not limited to nasal sprays, sinus rinses), over-the-counter medications (including but not limited to aspirin, decongestants, antihistamines, and other nonsteroidal anti-inflammatory drugs), and herbal medications (including but not limited to herbal tea or St. John s Wort) within 14 days prior to study enrollment, and agrees not to use these mediations through the final study visit, unless approved by the investigator.
  * Agrees not to donate blood or blood products from 3 months prior to enrollment through the final study visit.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Presence of self-reported or medically documented significant medical condition including but not limited to:

  * Chronic pulmonary disease (e.g., asthma, emphysema).
  * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
  * Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
  * Immunosuppression, immune deficiency, or ongoing malignancy.
  * Neurological and neurodevelopmental conditions (e.g., Bell s palsy, cerebral palsy, epilepsy, stroke, seizures).
  * Postinfectious or postvaccine neurological sequelae including GBS.
  * Body mass index (BMI) <= 18 and >= 35.
* Acute illness within 7 days prior to enrollment.
* Individuals who have grade 2 or above clinically significant laboratory values outside the limits thus specified by normal laboratory parameters.
* Known allergy to influenza vaccination or excipients contained in the influenza vaccine used.
* Known allergy to lidocaine or phenylephrine.
* Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
* Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
* Receipt of any unlicensed vaccine within 6 months prior to enrollment, not including COVID-19 vaccines under Emergency Use Authorization.
* Self-reported or known history of alcoholism or drug abuse within 6 months prior to enrollment, or positive urine test for drugs of abuse (i.e., amphetamines, cocaine metabolites, benzodiazepines, opiates, or tetrahydrocannabinol) prior to vaccination on V1D0.
* Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the principal investigator (PI) to be a contraindication to protocol participation.
* History of angioedema or anaphylaxis.
* History of SARS-COV-2 infection with residual or ongoing symptoms.
* Any condition or event that, in the judgment of the PI, is a contraindication to protocol participation or impairs the participant s ability to give informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2025-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.We are not working with any outside collaborators that require this information.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000320-I.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified and recruited from the community through multiple methodologies including local advertisement, direct contact of prior study participants, and word of mouth advertisement. Seventy-eight participants were screened between May 2022 and October 2022 on a separate screening protocol (11-I-0183).
Pre-assignment Details: Forty-five participants were enrolled and randomized to the three study arms.
Groups:
- Group A: 15 participants receiving IM BPL1357 and IN Placebo
- Group B: 15 participants receiving IN BPL1357 and IM Placebo
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 15 | 15 | 15
Received Dose 1 | 15 | 15 | 15
Received Dose 2 | 15 | 15 | 14 (One participant in the placebo group received their second vaccine late due to COVID-19. Another participant in the placebo group did not receive their second vaccine due to development of COVID-19 and subsequent schedule conflicts.)
Completed | 15 (One participant in the IM group missed their visit 28 days after the second dose of vaccine, when the primary immunogenicity analyses were performed) | 15 (One participant in the IN group withdrew consent after study completion. Safety data but not immunogenicity data are available for this participant.) | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.4) | 30.3 (10.2) | 27.5 (6.0) | 30.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 8 | 27
  Male | 3 | 8 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 13 | 14 | 15 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 10 | 7 | 9 | 26
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety - Serious Adverse Event
Description: Type of SAEs through day V2D28.
Time Frame: V2D28 (Day 56)
Measure: Number; unit: SAEs
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 15 | 15
SAEs | 0 | 0 | 0

2. Primary Outcome: Safety - Adverse Events
Description: Type and severity (by grading) of intervention-related AEs through day V2D28.
Time Frame: V2D28 (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Fatigue | 10 | 8 | 9
  Injection Site Pain | 14 | 6 | 0
  Headache | 8 | 3 | 6
  Myalgia | 4 | 3 | 2
  Sore Throat | 3 | 2 | 4
  Sneezing | 1 | 1 | 4
  Arthralgia | 1 | 3 | 1
  Hoarseness | 1 | 3 | 1
  Rhinorrhea | 1 | 2 | 2
  Nasal congestion | 0 | 1 | 3
  Neutrophil count decreased | 2 | 0 | 2
  Chills | 0 | 0 | 3
  Cough | 0 | 1 | 2
  Hypokalemia | 0 | 2 | 1
  Nausea | 1 | 1 | 1
  Decreased appetite | 0 | 0 | 2
  Hemoglobin decreased | 0 | 1 | 1
  Alanine aminotransferase increased | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 1
  Diarrhea | 0 | 1 | 0
  Dizziness | 0 | 1 | 0
  Erythema | 0 | 1 | 0
  Eye discomfort | 0 | 1 | 0
  Fever | 0 | 1 | 0
  Hyperglycemia | 1 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0
  Injection site ecchymosis | 1 | 0 | 0
  Migraine | 1 | 0 | 0
  Muscle weakness lower limb | 0 | 1 | 0
  Numbness | 1 | 0 | 0
  Pain | 0 | 1 | 0
  Paresthesia | 1 | 0 | 0
  Pruritus | 0 | 1 | 0
  Vertigo | 0 | 1 | 0
  WBC decreased | 1 | 0 | 0
  WBC increased | 0 | 0 | 1

3. Secondary Outcome: Safety - Serious Adverse Event
Description: Type of SAEs through day V2D182
Time Frame: V2D182 (Day 210)
Measure: Number; unit: SAEs
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 15 | 15
SAEs | 0 | 0 | 0

4. Secondary Outcome: Safety - Adverse Events
Description: Type and severity (by grading) of AEs through day V2D182
Time Frame: V2D182 (Day 210)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Fatigue | 10 | 8 | 9
  Injection site pain | 14 | 6 | 0
  Headache | 8 | 3 | 6
  Myalgia | 4 | 3 | 2
  Sore throat | 3 | 2 | 4
  Sneezing | 1 | 1 | 4
  Arthralgia | 1 | 3 | 1
  Hoarseness | 1 | 3 | 1
  Rhinorrhea | 1 | 2 | 2
  Nasal congestion | 0 | 1 | 3
  Neutrophil count decreased | 2 | 0 | 2
  Chills | 0 | 0 | 3
  Cough | 0 | 1 | 2
  Hypokalemia | 0 | 2 | 1
  Nausea | 1 | 1 | 1
  Decreased appetite | 0 | 0 | 2
  Hemoglobin decreased | 0 | 1 | 1
  Alanine aminotransferase increased | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 1
  Diarrhea | 0 | 1 | 0
  Dizziness | 0 | 1 | 0
  Erythema | 0 | 1 | 0
  Eye discomfort | 0 | 1 | 0
  Fever | 0 | 1 | 0
  Hyperglycemia | 1 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0
  Injection site ecchymosis | 1 | 0 | 0
  Migraine | 1 | 0 | 0
  Muscle weakness lower limb | 0 | 1 | 0
  Numbness | 1 | 0 | 0
  Pain | 0 | 1 | 0
  Paresthesia | 1 | 0 | 0
  Pruritus | 0 | 1 | 0
  Vertigo | 0 | 1 | 0
  WBC decreased | 1 | 0 | 0
  WBC increased | 0 | 0 | 1

5. Secondary Outcome: Immunogenicity - Systemic and Mucosal Immune Responses Against Hemagglutinin
Description: Antibodies against H1, H3, H5, and H7 head and stalk as measured by HAI or ELISA from blood and mucosal samples at V2D28
Time Frame: V2D28 (Day 56)
Population: One participant in Group A missed their V2D28 visit and did not provide samples for analysis at this timepoints. One participant in group B withdrew consent to use samples after study completion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Titers
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 15
ELISA Titers
  Serum Anti-H1 IgG | 2765 (4339) [1580 to 4839] | 2093 (2519) [1309 to 3345] | 1776 (1514) [1223 to 2580]
  Serum Anti-H3 IgG | 1104 (973) [737 to 1653] | 379 (686) [202 to 710] | 333 (242) [219 to 505]
  Serum Anti-H5 IgG | 1010 (1425) [632 to 1615] | 365 (310) [234 to 569] | 284 (145) [210 to 386]
  Serum Anti-H7 IgG | 638 (524) [452 to 902] | 169 (421) [92 to 311] | 141 (123) [86 to 231]
  Nasal Anti-H1 IgA | 0.446 (0.520) [0.288 to 0.690] | 0.556 (0.325) [0.411 to 0.754] | 0.504 (0.223) [0.375 to 0.676]
  Nasal Anti-H3 IgA | 0.525 (0.218) [0.420 to 0.655] | 0.564 (0.279) [0.438 to 0.726] | 0.543 (0.267) [0.418 to 0.706]
  Nasal Anti-H5 IgA | 0.213 (0.332) [0.132 to 0.343] | 0.377 (0.345) [0.242 to 0.589] | 0.264 (0.291) [0.168 to 0.415]
  Nasal Anti-H7 IgA | 0.279 (0.316) [0.185 to 0.421] | 0.357 (0.131) [0.285 to 0.446] | 0.329 (0.210) [0.236 to 0.460]

6. Secondary Outcome: Immunogenicity - Systemic and Mucosal Immune Responses Against Neuraminidase
Description: Antibodies against N1, N3, N8, and N9 as measured by NAI or ELISA from blood and mucosal samples at V2D28
Time Frame: V2D28 (Day 56)
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Titers
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 15
ELISA Titers
  Serum Anti-N1 IgG | 222 [119 to 415] | 266 [138 to 513] | 282 [184 to 432]
  Serum Anti-N3 IgG | 43 [19 to 100] | 30 [17 to 52] | 20 [13 to 29]
  Serum Anti-N8 IgG | 25 [15 to 44] | 15 [10 to 22] | 23 [13 to 41]
  Serum Anti-N9 IgG | 25 [13 to 46] | 12 [10 to 16] | 13 [10 to 17]
  Nasal Anti-N1 IgA | 0.171 [0.111 to 0.264] | 0.405 [0.264 to 0.622] | 0.308 [0.169 to 0.561]
  Nasal Anti-N3 IgA | 0.091 [0.076 to 0.110] | 0.132 [0.091 to 0.190] | 0.142 [0.089 to 0.226]
  Nasal Anti-N8 IgA | 0.139 [0.102 to 0.190] | 0.238 [0.165 to 0.343] | 0.288 [0.178 to 0.464]
  Nasal Anti-N9 IgA | 0.124 [0.095 to 0.162] | 0.164 [0.164 to 0.252] | 0.240 [0.152 to 0.379]

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=15) | Group B (N=15) | Group C (N=15)
Fatigue (General disorders) | 12 | 9 | 10
Injection site pain (General disorders) | 15 | 6 | 6
Headache (Nervous system disorders) | 10 | 7 | 9
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 10
Respiratory rate (Investigations) | 5 | 10 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 8 | 5
Bradycardia (Investigations) | 4 | 5 | 5
Hypokalemia (Metabolism and nutrition disorders) | 3 | 5 | 6
Hemoglobin decreased (Investigations) | 6 | 3 | 4
CPK increased (Investigations) | 2 | 5 | 5
Neutrophil count decreased (Investigations) | 3 | 3 | 6
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4
Chills (General disorders) | 3 | 4 | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6
COVID-19 (Infections and infestations) | 3 | 1 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 4
Upper respiratory infection (Infections and infestations) | 4 | 2 | 1
Fever (General disorders) | 1 | 3 | 2
Hyponatremia (Investigations) | 2 | 3 | 1
Hypophosphatemia (Investigations) | 2 | 0 | 4
Lymphocyte count decreased (Investigations) | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal cramps (Gastrointestinal disorders) | 3 | 0 | 1
WBC decreased (Investigations) | 1 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 2
Eye discomfort (Eye disorders) | 0 | 2 | 1
Feverish (General disorders) | 2 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
WBC increased (Investigations) | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rhinovirus infection (Investigations) | 0 | 1 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Anterior cruciate ligament tear (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BUN increased (Investigations) | 0 | 1 | 0
Cotton wool spots (Eye disorders) | 1 | 0 | 0
Dental implant user (Social circumstances) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Difficulty thinking (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Injection site ecchymosis (General disorders) | 1 | 0 | 0
Injection site itching (General disorders) | 0 | 0 | 1
Itchy throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Loss of smell (Nervous system disorders) | 0 | 0 | 1
Low back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Meniscus tear of knee (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Menstrual irregularity (Reproductive system and breast disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Numbness (Nervous system disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Puncture wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Smell alteration (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Systolic hypertension (Vascular disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Taste alteration (Nervous system disorders) | 1 | 0 | 0
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Uric acid high (Investigations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Venipuncture site bruise (General disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Weight loss (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05027932/Prot_SAP_000.pdf